CLINICAL TRIAL: NCT02719613
Title: Continuing Treatment for Subjects Who Have Participated in a Prior Protocol Investigating Elotuzumab
Brief Title: Continuing Treatment for Participants Who Have Participated in a Prior Protocol Investigating Elotuzumab
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CA204-185; 2016-000037-51 (EudraCT Number)
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Dexamethasone; Lenalidomide; Bortezomib; pomalidomide; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elotuzumab (Experimental): This is a continuation roll-over study for patients receiving benefit from prior elotuzumab protocols. All participants will receive elotuzumab and/or other study drugs as per previous protocol.
  Interventions: Drug: Elotuzumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Bortezomib; Drug: Pomalidomide; Drug: Nivolumab

INTERVENTIONS:
Drug: Elotuzumab — Patients will continue to receive treatment with the investigational study drug by intravenous (IV) solution administration at the last dose and schedule received in the previous study.
  Other Names: BMS-901608; HuLuc63; Empliciti
Drug: Dexamethasone — Patients will continue to receive treatment with non-investigational study drug by oral tablet administration at the last dose and schedule received in the previous study.
Drug: Dexamethasone — Patients will continue to receive treatment with non-investigational study drug by intravenous (IV) solution administration at the last dose and schedule received in the previous study.
Drug: Lenalidomide — Patients will continue to receive treatment with non-investigational study drug by oral capsule administration at the last dose and schedule received in the previous study.
  Other Names: Revlimid®
Drug: Bortezomib — Patients will continue to receive treatment with non-investigational study drug by intravenous (IV) or subcutaneous injection solution administration at the last dose and schedule received in the previous study.
  Other Names: Velcade®
Drug: Pomalidomide — Patients will continue to receive treatment with non-investigational study drug by oral capsule administration at the last dose and schedule received in the previous study.
  Other Names: Pomalyst ®
Drug: Nivolumab — Patients will continue to receive treatment with the investigational study drug by intravenous (IV) solution administration at the last dose and schedule received in the previous study.
  Other Names: Opdivo ®

SUMMARY:
The purpose of this study is to continue to provide elotuzumab and/or other study drugs to participants who have participated on a prior protocol investigating elotuzumab who are not able to receive commercial drug supply.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participated in a previous elotuzumab protocol (including, but not limited to HuLuc63-1703, CA204007, CA204009, or CA204011) and is deemed by the investigator to be deriving benefit from elotuzumab and/or other study drugs as defined by the previous protocol
* Receiving elotuzumab and/or other study drugs at the time of signature of informed consent
* Males and Females, ages 18 and older

Exclusion Criteria:

* All participants previously discontinued from an elotuzumab study for any reason
* Participants not receiving clinical benefit from previous study therapy
* Participants who are not medically well enough to receive study therapy as determined by the investigator

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
The number of participants who received at least one dose of elotuzumab or backbone therapy (other study drugs) and the duration of treatment will be collected. | Maximum duration is until all participants have discontinued study drugs, or until all participants are treated for up to 2 years, unless BMS chooses to extend the study.

SECONDARY OUTCOMES:
All serious adverse events (SAEs) will be collected. | Maximum duration is until all participants have discontinued study drugs, or until all participants are treated for up to 2 years, unless BMS chooses to extend the study.
All Grade 5 adverse events (AEs) will be collected. | Maximum duration is until all participants have discontinued study drugs, or until all participants are treated for up to 2 years, unless BMS chooses to extend the study.
All adverse events (AEs) previously not reported will be collected. | Maximum duration is until all participants have discontinued study drugs, or until all participants are treated for up to 2 years, unless BMS chooses to extend the study.
All adverse events (AEs) leading to discontinuation will be collected. | Maximum duration is until all participants have discontinued study drugs, or until all participants are treated for up to 2 years, unless BMS chooses to extend the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (41):
- United States (14):
  - Local Institution - 0020, Tucson, Arizona
  - Local Institution - 0017, Bakersfield, California
  - Local Institution - 0022, Fountain Valley, California
  - Local Institution - 0016, West Hollywood, California
  - Local Institution - 0019, Denver, Colorado
  - Local Institution - 0021, Jacksonville, Florida
  - Local Institution - 0042, St. Petersburg, Florida
  - Local Institution - 0009, Atlanta, Georgia
  - Local Institution - 0003, Indianapolis, Indiana
  - Local Institution - 0002, Boston, Massachusetts
  - Local Institution - 0008, St Louis, Missouri
  - Local Institution - 0004, New York, New York
  - Local Institution - 0001, Bethlehem, Pennsylvania
  - Local Institution - 0018, Dallas, Texas
- Local Institution - 0034, Heidelberg, Victoria, Australia
- Local Institution - 0023, Antwerp, Belgium
- Canada (2):
  - Local Institution - 0011, Toronto, Ontario
  - Local Institution - 0010, Halifax
- Local Institution - 0035, Athens, Greece
- Local Institution - 0036, Budapest, Hungary
- Italy (6):
  - Local Institution - 0015, Ancona
  - Local Institution - 0012, Florence
  - Local Institution - 0013, Genova
  - Local Institution - 0043, Ravenna
  - Local Institution - 0044, Terni
  - Local Institution - 0014, Torino
- Japan (6):
  - Local Institution - 0046, Aomori, Aomori
  - Local Institution - 0047, Shibukawa-shi, Gunma
  - Local Institution - 0049, Osaka, Osaka
  - Local Institution - 0048, Koto-ku, Tokyo
  - Local Institution - 0050, Chiba
  - Local Institution - 0045, Kasama-shi
- Poland (3):
  - Local Institution - 0027, Chorzów
  - Local Institution - 0026, Warsaw
  - Local Institution - 0039, Warsaw
- Romania (2):
  - Local Institution - 0028, Bucharest
  - Local Institution - 0029, Iași
- Spain (2):
  - Local Institution - 0041, Barcelona
  - Local Institution - 0030, Toledo
- Local Institution - 0031, Cebeci Ankara, Turkey (Türkiye)
- Local Institution - 0032, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT02719613.html